CLINICAL TRIAL: NCT04260503
Title: Analysis of Gut Microbiome and Liver Imaging Including Elasticity in Biliary Atresia Patients With Cholangitis for the Prediction of Disease Activity and Improvement of Outcome Using Fecal Microbiota Transplantation
Brief Title: Gut Microbiome in Biliary Atresia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0306
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Biliary Atresia
Keywords: Biliary atresia; Microbiota; Cholangitis
MeSH Terms: conditions — Biliary Atresia; Cholangitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Biliary Atresia: Disease group
  Interventions: Other: Monitoring of the gut-microbiome and ultrasound elasticity.
- Choledochal cyst: Disease control
  Interventions: Other: Monitoring of the gut-microbiome
- Neonatal hepatitis: Disease control
  Interventions: Other: Monitoring of the gut-microbiome
- Healthy baby: Healthy control
  Interventions: Other: Monitoring of the gut-microbiome.

INTERVENTIONS:
Other: Monitoring of the gut-microbiome and ultrasound elasticity. — The investigator will investigate the alteration of gut-microbiome and liver stiffness by restoration of bile flow by operation.
  Groups: Biliary Atresia
Other: Monitoring of the gut-microbiome — The investigator will investigate the alteration of gut-microbiome before and after operation.
  Groups: Choledochal cyst
Other: Monitoring of the gut-microbiome — The investigator will investigate the alteration of gut-microbiome along with the disease progress.
  Groups: Neonatal hepatitis
Other: Monitoring of the gut-microbiome. — The investigator will investigate the alteration of gut-microbiome according to the normal development.
  Groups: Healthy baby

SUMMARY:
The investigator will investigate the gut-microbiome and liver elasticity of the Biliary Atresia (BA)-patients before and after Kasai operation. The data will be analyzed according to their clinical outcomes including cholangitis to find out diagnostic makers, significantly associated with the BA-phenotypes. The decision-making tree for the BA will be updated with our data, which will strength the prognosis and prediction. The establishment of gut-liver axis, featured by cholangitis and gut-microbiome will open new pathway to treat the BA using fecal microbiota transplantation.

1. Analysis of gut-microbiome: The investigator will investigate the alteration of gut-microbiome by restoration of bile flow at diagnosis, before and after Kasai procedure. In case of cholangitis after Kasai operation, signature gut-microbiome will be analyzed, which will lead to prevention of BA-patients from cholangitis via the bacteria transplantation.
2. Analysis of elastography: In order to improve non-invasive diagnosis, The investigator will investigate the alteration of liver elasticity and hepatic blood flow before and after Kasai procedure as well as upon cholangitis and choledochal cyst. Those data will be analyzed in parallel with serum biochemical markers to be associated with pathophysiological events e.g., cholestasis, cholangitis and fibrosis.

ELIGIBILITY:
1. Biliary atresia (Disease)

   Inclusion Criteria:
   * 0-4 months old
   * Patients, diagnosed with the BA and scheduled for Kasai operation during our study period
   * Patients whose parents or guardian understand our research aims, and comply to participate in our researches

   Exclusion Criteria:
   * Patients, whose diagnosis of BA was not definite.
   * Patients, scheduled for Kasai operation after 4 months old
2. Choledochal cyst (Disease control)

   Inclusion Criteria:
   * 0-7 years old
   * Patients, diagnosed with choledochal cyst and scheduled for total cyst removal during our study period
   * Patients whose parents or guardian understand our research aims, and comply to participate in our researches

   Exclusion Criteria:
   * Patients, whose diagnosis of choledochal cysts was not definite.
   * Patients with choledochal cyst, but greater than 7 years old
3. Neonatal hepatitis (Disease control)

   Inclusion Criteria:
   * 0-4 months old
   * Patients, diagnosed with the neonatal hepatitis during our study period
   * Patients whose parents or guardian understand our research aims, and comply to participate in our researches

   Exclusion Criteria:
   * Patients with hepatobiliary infection
   * Patients, required to use antibiotics to treat the infection
   * Patients with hepatobiliary inflammation, caused by abnormal intra- or extra-hepatic structure
4. Healthy control

Inclusion Criteria:

* 0-4 months old
* Healthy neonates without chronic diseases when they visit for vaccination
* Healthy neonates whose parents or guardian understand our research aims, and comply to participate in our researches

Exclusion Criteria:

* Patients with hepatobiliary infection
* Patients, required to use antibiotics to treat the infection
* Neonates with less than 37 weeks (i.e., preterm) or hospitalized in neonatal intensive care unit
* Patients, diagnosed with congenital malformation, syndrome and chronic diseases

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Biliary atresia Patients, diagnosed with the BA and scheduled for Kasai operation at Severance children's hospital during study period
  2. Choledochal cyst Patients, diagnosed with choledochal cyst and scheduled for total cyst removal at Severance children's hospital during study period
  3. Neonatal hepatitis Patients, diagnosed with the neonatal hepatitis during study period at Severance chilren's hospital
  4. Healthy control Healthy neonates without chronic diseases when they visit Severance chilren's hospital for vaccination
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
The changes of gut-microbiome according to the disease. | 1year
  Using shotgun metagenomic analysis, we will analyze the alteration of gut-microbiota according to the disease phenotypes.

SECONDARY OUTCOMES:
Comparison of gut microbiome according to the clinical outcomes of biliary atresia. | 1year
  The investigator will compare gut-microbiome according to the disease prognosis measured by ultrasound elastography and laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Gastroenterology, Hepatology and Nutrition, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided